CLINICAL TRIAL: NCT01832467
Title: A Pilot Case-control Study of Second or Third Line Treatment With Cetuximab-containing Chemotherapy in Patients With Metastatic Colorectal Cancer Who Were Previously Treated With Cetuximab-based Chemotherapy
Brief Title: Cetuximab Rechallenge Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COL019
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: cetuximab-based chemotherapy; previously treated
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cetuximab-containing chemotherapy (Experimental): * Cetuximab may be given at either one of the following schedules at the investigator's discretion:
    1. 2-weekly: Cetuximab is started on day 1 of each cycle of chemotherapy, at 500mg/m2 every 2 weeks over 120/90/60minutes.
    2. Weekly: Cetuximab may be given at a loading dose of 400mg/m2 on day 1over 120 minutes, followed by weekly dosing at 250mg/m2 on day 1, over 60 minutes of each cycle of chemotherapy.
  * Chemotherapy: Only one of the following regimens may be combined with cetuximab at the investigator's discretion according to institutional standard. Some recommended regimens used in Hong Kong.
  Regimens to be combined with biweekly cetuximab:
  1. Irinotecan at 2-weekly schedule.
  2. FOLFIRI (as inpatient or via ambulatory pump).
  3. FOLFOX (as inpatient or via ambulatory pump).
  Interventions: Drug: cetuximab-containing chemotherapy

INTERVENTIONS:
Drug: cetuximab-containing chemotherapy

SUMMARY:
To determine the objective overall response of re-treatment with cetuximab-based chemotherapy in patients upon disease progression while under observation, who had previously responded to first-line or second-line treatment with cetuximab-based chemotherapy for metastatic colorectal cancer (mCRC), but had stopped treatment for reasons other than disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Able to give written informed consent.
* Histologically confirmed colorectal adenocarcinoma: must be either metastatic disease or unresectable recurrent disease.
* KRAS mutation status of the primary or metastastic CRC tumor must be wild-type.
* ECOG performance status of 0-1 at study entry.
* Must have measurable disease by RECIST (ver 1.1) criteria.
* Have progressive disease based on all of the following criteria (from a-d):

  (a) Previously received cetuximab-based chemotherapy as first- or second-line treatment for metastatic or recurrent disease with, any one of the following drug combinations: (i) Cetuximab, fluoropyrimidines and oxaliplatin; or, (ii) Cetuximab, fluoropyrimidines and irinotecan; or (iii) Cetuximab and irinotecan. (b) Must have achieved at least stable disease, partial or complete response to treatment stated in '(a)' above.

  (c) Experienced disease progression after more than 60 days from the last date of administration of the treatment stated in '(a)' above.

  (d) 'Disease progression' can be defined as radiological or clinical progression.
* Adequate hematologic, renal, hepatic function as defined by: absolute neutrophil count >= 1.5 x 109/L, hemoglobin >= 9 g/L, platelets >= 100 x 109/L, calculated creatinine clearance >=55 ml/min, total bilirubin <= 2 x the upper limit of normal (ULN), alanine aminotransferase (ALT) <2.5 upper limit of normal or <= 5 x ULN in the presence of liver metastases.
* Must have recovered to grade 0-1 in severity, any toxicity related to previous cetuximab.

Exclusion Criteria:

* Disease progression during first-line or second-line treatment with cetuximab and chemotherapy in combination.
* Patients who had prior cetuximab in BOTH first and second-line setting.
* Previous use of bevacizumab.
* Prior grade 3 to 4 hypersensitivity reaction to cetuximab.
* Clinically significant and poorly controlled medical illnesses within the last 6 months which may be exacerbated by study treatment.
* Estimated life expectancy of less than 3 months.
* Radiotherapy, surgery (excluding prior diagnostic biopsy) or any investigational drug in the 30 days before enrollment. Radiotherapy for pain relief is allowed as long as not targeted at an index or non-index lesion, e.g., bone metastases.
* Known brain and/or leptomeningeal metastases.
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction within the last twelve months, significant arrhythmias
* Pregnancy or lactation
* Previous malignancy other than colorectal cancer in the last 5 years except basal cell cancer of the skin or preinvasive cancer of the cervix. The non-CRC malignancy must be in known complete remission for at least 5 years prior to enrollment.
* The presence of KRAS mutation in any of the CRC tumor tissue(s) - for example, patients with synchronous primary CRCs with different KRAS mutation status.
* Participants with reproductive potential who are unwilling to perform effective contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-04-24; Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
overall response of re-treatment with cetuximab-based chemotherapy | 2 years
  in patients experiencing disease progression while under observation, who had previously responded to first-line or second-line treatment with cetuximab-based chemotherapy for metastatic colorectal cancer (mCRC), but had stopped treatment for reasons other than disease progression.

SECONDARY OUTCOMES:
Adverst event and toxicity during treatment period | 2 years
disease control rate | 2 years
progression-free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Brigette MA, MD, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong